CLINICAL TRIAL: NCT06979440
Title: Study on the Molecular Mechanism of Berberine Regulating the Gut Microbiota-derived Metabolites 5-AVAB to Improve Type 2 Diabetes Mellitus Complicated With Depression.
Brief Title: Study on the Molecular Mechanism of Berberine to Improve Type 2 Diabetes Mellitus Complicated With Depression
Acronym: SBDD
Status: Recruiting | Type: Observational
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-K231-01; 82404740 (Other Grant/Funding Number: National Natural Science Foundation of China); 202495102 (Other Grant/Funding Number: Jiangsu Pharmaceutical Association)
Record Dates: First submitted 2025-05-13; First posted 2025-05-20 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-01

CONDITIONS: Diabetes-Related Complications
Keywords: Type 2 diabetes mellitus; depression; Diabetes Complications
MeSH Terms: conditions — Diabetes Complications; Diabetes Mellitus, Type 2; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — faeces and blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control (with type 2 diabetes): The clinical inclusion criteria are as follows:
  a. Age 18-65 years old; b. The Con group was diagnosed with type 2 diabetes and had no history of mental disorders such as depression; c. No antibiotics, prebiotics, probiotics, enteral nutrition drugs, etc. were used within 3 months before diagnosis, and no antibiotics, prebiotics, probiotics, enteral nutrition drugs, etc. were used during treatment.
  Interventions: Other: No intervention
- T2DD (with type 2 diabetes complicated with depression): The clinical inclusion criteria are as follows:
  a. Age 18-65 years old; b. The T2DD patient group was diagnosed with type 2 diabetes complicated with depression (depression met the DSM-5 diagnostic criteria); c. No antibiotics, prebiotics, probiotics, enteral nutrition drugs, etc. were used within 3 months before diagnosis, and no antibiotics, prebiotics, probiotics, enteral nutrition drugs, etc. were used during treatment.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The incidence of type 2 diabetes with comorbid depression (T2DD) is notably high, characterized by prolonged disease duration and susceptibility to recurrence. The preliminary experiments identified 5-AVAB, a gut microbiota-derived metabolite, as a potential novel biomarker for T2DD progression. Given the absence of existing research in this area, it warrants in-depth investigation.

The investigators plan to collect fecal and serum samples from participants with type 2 diabetes and those with T2DD to quantify 5-AVAB levels, as well as conduct in vitro gut microbiota culturing and sequencing studies.

DETAILED DESCRIPTION:
This study will enroll two groups of participants: a control group (with type 2 diabetes) and a T2DD group (with type 2 diabetes with comorbid depression) (n=20 per group). From each participant, 5 mL of whole blood and 5 g of fresh stool will be collected. The whole blood samples will be processed for serum extraction. The 5-AVAB concentrations in all samples will be quantified using LC-MS/MS and compared between groups.

Anaerobic culture medium will be prepared, and the fresh stool samples will be homogenized with the medium at a ratio of 1 g:20 mL. After 20 minutes of pre-incubation at 37°C under anaerobic conditions, berberine will be added at concentrations of 10 μg/mL, 50 μg/mL, and 100 μg/mL, followed by incubation for 2, 6, 12, and 24 hours. The 5-AVAB levels in each group will then be measured using LC-MS/MS. The additional requirements are as follows:

1. Exit and termination criteria If the subject stops the study before sampling, it will be regarded as exit/termination of the study.
2. The time the participants participated in the study (each time and total time) The time from the start of the group to the completion of sampling is regarded as the time of participation in the study.
3. Recruitment process After review and approval by the Ethics Committee of the Affiliated Hospital of Nantong University, this study can start recruiting. It is planned to recruit in the Department of Endocrinology and Department of Neurology of this hospital, and it is expected to recruit 40 participants without any compensation.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-65 years (including the critical value), regardless of gender;
2. The Con group was diagnosed with type 2 diabetes and had no history of mental disorders such as depression;
3. The T2DD patient group was diagnosed with type 2 diabetes and depression, where depression met the DSM-5 diagnostic criteria for recurrent depression without psychotic symptoms or single-episode MDD, and the total score of the HAMD-17 scale was ≥22 points;
4. The subjects read and fully understood the patient instructions and signed the informed consent form.

Exclusion Criteria:

1. Those who do not meet the inclusion criteria;
2. Those who have not used antibiotics, prebiotics, probiotics, enteral nutrition drugs, etc. within 3 months before diagnosis, and those who do not use antibiotics, prebiotics, probiotics, enteral nutrition drugs, etc. during treatment;
3. Those with progressive serious diseases (such as cancer);
4. Those with severe aphasia, agnosia, and apraxia;
5. Those who have used psychotropic drugs for a long time within 1 month before the study or have received new drug research in the past 3 months;
6. Pregnant or breastfeeding women;
7. Alcoholics or drug addicts;
8. Those with poor mental condition and unable to cooperate;
9. Those who are considered unsuitable for inclusion in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Con group was diagnosed with type 2 diabetes and had no history of mental disorders such as depression; The T2DD patient group was diagnosed with type 2 diabetes and depression, where the depression met the DSM-5 diagnostic criteria for recurrent depression without psychotic symptoms or single-episode MDD, and the total score of the HAMD-17 scale was ≥22 points;
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-11-09 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The levels of 5-AVAB | 3 years
  There were no additional intervention measures in this study. Faeces were collected after excretion for in vitro drug intervention experiments. The blood collection volume (5 mL) met the ISO international standard and was used to detect the 5-AVAB content in each group.

CONTACTS AND LOCATIONS:
Overall Officials: zhengwei zhang, PhD, Principal Investigator — Affiliated Hospital of Nantong University
Locations (1):
- Affiliated Hospital of Nantong University, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-05-18): https://cdn.clinicaltrials.gov/large-docs/40/NCT06979440/Prot_SAP_000.pdf
  • Informed Consent Form (2025-05-18): https://cdn.clinicaltrials.gov/large-docs/40/NCT06979440/ICF_001.pdf